CLINICAL TRIAL: NCT04364360
Title: Fatty Acid MetabOlism in Individuals Undergoing Sulforaphane Supplementation (FAMOUS)
Brief Title: Sulforaphane Supplementation Study
Acronym: FAMOUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Quadram Institute Bioscience (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1439
Record Dates: First submitted 2020-04-06; First posted 2020-04-28 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Obesity; Metabolic Syndrome
Keywords: Sulforaphane; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Metabolic Syndrome | interventions — sulforaphane

STUDY DESIGN:
Intervention Model Description: Single group intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sulforaphane supplementation (Experimental): Daily (2 capsules) consumption of BroccoMax (Jarrow Formulas Los Angeles, CA) for 3-weeks.
  Interventions: Dietary Supplement: Sulforaphane extract

INTERVENTIONS:
Dietary Supplement: Sulforaphane extract — 2x BroccoMax® capsules day, giving a total daily dose of 30 mg of Sulforaphane Glucosinolate Per day

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is increasing in the population, and is associated with heart disease and diabetes. At present there are no licensed drugs for treatment of NAFLD, therefore changes in diet and increased physical activity leading to decreased body fatness is the recommended management/treatment strategy. However, these are difficult to achieve and maintain for many individuals. A potential compound gaining interest in regards the treatment/prevention of NAFLD is sulforaphane, which is found in vegetables such as Broccoli. Animal studies suggest supplementing with sulforaphane can increase fat oxidation. This increased "fat burning" may result in lower levels of fat in the liver and overall in the body.

The researchers will ask participants to undertake an intervention phase which will involve consuming two sulforaphane tablets a day for approximately 3 weeks. Participants will be asked to maintain all other aspects of their lifestyle throughout the intervention phase. The researchers will measure and compare participants whole-body and liver fat oxidation in response to a standardised test meal before and after the intervention phase by taking blood and breath samples. The researchers will also measure the amount of fat in participants liver and heart using a non-invasive technique known as magnetic resonance spectroscopy (MRS) before and after the intervention.

DETAILED DESCRIPTION:
Participants satisfying the inclusion criteria will be invited to the Oxford Centre for Clinical Magnetic Resonance Research (OCMR), to measure the amount of fat within their liver and heart using magnetic resonance imaging and spectroscopy (MRI/S). Then on a separate day, within one week of having their liver and heart fat content measured, participants will come into the Clinical Research Unit (CRU) at the Oxford Centre for Diabetes Endocrinology and Metabolism (OCDEM) for a 'postprandial study day' after an overnight fast. Participants will be asked to avoid excessive exercise and alcohol for 24 hours prior to the study. The day prior to and over the course of the 'study day' participants will be asked to drink some 'heavy water' ((2H2O) CK Isotopes Limited). The amount of 'heavy water' a volunteer will have to consume is 3g heavy water per kg body water, which will achieve a plasma water enrichment of 0.3%. Once participants arrive at OCDEM the researchers will make some anthropometric measurements (e.g. weight, height, waist circumference etc.), collect a urine sample, and place a small plastic tube (cannula) into a vein on the forearm, from which they will take blood samples. A second cannula will also be placed into a large vein in the elbow crease of the opposite arm. Sequential blood samples will be collected by the researchers at regular intervals for a period of up to 8 hours from placing the first cannula. After the first blood samples have been taken (Time -30) the researchers will start pumping fat labelled with special atoms (stable isotopes from CK Isotopes Limited) into the other cannula. After approximately 30 minutes of infusion, a second blood sample (time 0) will be taken, after which participants will be fed a standardised test meal which will consist of cereal and semi-skimmed milk and a "fatty" chocolate drink. The fatty chocolate drink is made with a blend of oils and will be labelled with a stable isotope (from CK Isotopes Limited). The use of the stable isotopes in small doses is considered to be completely harmless (it is not radioactive). Once the test meal is consumed, the volunteer is free to rest on a bed or in a chair, as they prefer, until the experiment is finished, up to 8 hours. After giving the stable isotopes, blood and breath samples will be taken initially every 30 minutes for the first two hours and then every 60 minutes up until the end of the study day (6 hours post breakfast). The researchers would take blood samples through the cannula in the vein, and at each time point would take approx. 25ml of blood. The most blood taken in total over the day would be 250ml or approximately 1/2 of a pint.

Three hours after consumption of the test breakfast meal the researchers will take two adipose tissue biopsies. The first biopsy will be taken from the fat just under the skin in the abdomen (tummy) and the second biopsy will be taken from the gluteal (buttock) region. There will be numbing of the skin and fat tissue as a local anaesthetic (1% lignocaine) is used prior to all biopsies. The choice as to whether or not to undergo biopsies will be given to participants on the study day. At some point during the day a dual energy X-ray absorptiometry (DEXA) scan will be performed. The DEXA scan will measure the total amount of fat (adipose tissue) along with the amount of adipose tissue in specific depots (e.g. upper body, lower body, visceral etc.). When all of the samples have been taken and the measurements are finished, the researchers would take out the plastic tubes, and give the participant something further to eat and drink before making sure they can get home, usually by providing them with a taxi. Participants will also be provided with the sulforaphane capsules to be ingested over the following 3-week period, and guidelines as to when to take supplements. Participants will be asked to maintain their habitual diets during the intervention phase, which will be assessed via the completion of food diaries where all foods and beverages consumed on 3 days a week (two week and one weekend day) each week of the 3 week intervention phase. A member of the research team will be in regular contact with participants via email throughout the intervention phase in an attempt to maintain compliance. Following the 3-week intervention phase the volunteer's liver and heart fat content will again be measured using MRI/S at OCMR, then on a separate day, within one week of having their liver and heart fat content measured, participants will come into the CRU at OCDEM for a second 'study day' after an overnight fast. The second 'study day' will be identical to the first study day described above.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Healthy adults, Male or Female, aged 18 to 65 years.
* No medical condition or relevant drug therapy known to affect glucose or fatty acid metabolism.
* Weight stable for the previous 3 months. -

Exclusion Criteria:

* Aged ≤18 or ≥65 years.
* Body Mass Index ≤19 or ≥35kg/m2.
* Females with a body mass ≤50kg.
* A blood haemoglobin <135mg/dL for men and <120mg/dL for women.
* Donated (or lost) ≥250 ml of blood in the previous two months.
* On a weight loss diet or have decreased their body weight by >5% in the previous 3 months.
* Have increased their body weight by >5% in the previous 3 months.
* Any metabolic condition or relevant drug therapy known to affect glucose or fatty acid metabolism.
* Smoking, or use of nicotine replacement agents (e.g. e-cigarettes).
* History of alcoholism or a greater than recommended alcohol intake (>30 g of alcohol daily for men and >20 g of alcohol daily for women).
* Current or history of Haemorrhagic disorders.
* History of albumin allergy or allergic to eggs
* Current or history of anticoagulant treatment.
* Pregnant or nursing mothers.
* Women prescribed any hormone replacement therapy (HRT) or who have used these within the last 12 months.
* History of severe claustrophobia.
* Presence of metallic implants, pacemaker, or inability/unwillingness to remove any piercings, and any large tattoos around the area to be scanned.
* History or current psychiatric illness.
* History or current neurological condition (e.g. epilepsy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Change in whole-body fatty acid oxidation | within 7 days after completion of the intervention
  Stable-isotope tracers will be used to measure whole-body dietary fatty acid oxidation in response to a standardised test meal before and after the intervention.

SECONDARY OUTCOMES:
Change in liver fat content | within 7 days after completion of the intervention
  MRI/S will be used to measures liver fat content before and after the intervention.
Change in hepatic fatty acid partitioning | within 7 days after completion of the intervention
  Stable-isotope tracers will be used to measure whole-body and hepatic fatty acid metabolism in response to a standardised test meal before and after the intervention.
Change in glycemic control | within 7 days after completion of the intervention
  Participants postprandial glycemic control will be measured following a standardised test meal before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Hodson, PhD, Principal Investigator — University of Oxford
Locations (1):
- Oxford Centre for Diabetes, Endocrinology and Metabolism, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No